CLINICAL TRIAL: NCT05753085
Title: Multimodality Optical and Ultrasound Intravascular Imaging for Stent Optimization and Atheroma Assessment
Acronym: MOUSA
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Concerns with capacity
Sponsor: Barts & The London NHS Trust (Other)
Collaborators: Rosetrees Trust (Other); National Institute for Health Research, United Kingdom (Other Government); Conavi Medical Inc (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 268761
Record Dates: First submitted 2023-01-12; First posted 2023-03-03 (Actual); Last update posted 2025-09-17 (Actual); Status verified 2025-09

CONDITIONS: Coronary Artery Disease; Coronary Stenosis; Plaque, Atherosclerotic
Keywords: Coronary; Intravascular Imaging; Plaque
MeSH Terms: conditions — Coronary Artery Disease; Coronary Stenosis; Plaque, Atherosclerotic; Plaque, Amyloid | interventions — Tomography, Optical Coherence

STUDY DESIGN:
Intervention Model Description: A single-centre, prospective, non-randomized, open-label feasibility study of the Conavi Medical Novasight Hybrid System (IVUS and OCT) for stent optimization and atheroma assessment in patients who present with non-ST elevation myocardial infarction (NSTEMI).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Conavi Medical Novasight Hybrid System intervention (Experimental): Patients who present with non-ST elevation myocardial infarction (NSTEMI) and require an angiogram and or PCI will have intravascular imaging assessment of the culprit vessel using the Conavi Medical Hybrid System (Novasight Hybrid Catheter, Novasight Hybrid PIM, Novasight Hybrid Hummingbird Console)
  Interventions: Device: Conavi Medical Novasight Hybrid System intervention

INTERVENTIONS:
Device: Conavi Medical Novasight Hybrid System intervention — Patients for a coronary angiogram who meet the inclusion criteria and none of the exclusion criteria are enrolled. Participants are prepared for angiography and PCI procedure in the usual way. Radial or femoral artery cannulation is done under local anaesthetic and the angiogram performed as per standard practice. IVUS-OCT imaging of the culprit vessel using the Novasight Hybrid system is then performed. If image quality of the IVUS-OCT is suboptimal it will be repeated. If the IVUS-OCT catheter cannot cross the lesion, pre-dilatation is performed. The acquired IVUS-OCT images can be used to optimise PCI. Following PCI, angiography is repeated and if the findings are optimal, IVUS-OCT imaging is repeated. If the PCI results are suboptimal further stent optimisation is performed and IVUS-OCT imaging repeated; The procedure is then completed as clinically indicated. The participant will then receive conventional post PCI care
  Other Names: IVUS & OCT

SUMMARY:
This investigation is to see if the new Novasight Hybrid imaging catheter can safely and accurately provide two different types of images (IVUS and OCT) of the inside of heart vessels at the same time. The images will be compared against one type of image (IVUS) to see if providing two, improves identification of different types of plaque (fatty substances) and informs better treatment.

Atherosclerotic coronary artery disease is the name given to the development of plaques in the heart vessels. The plaques can cause narrowing in the vessels which may cause chest pain. Sometimes, plaques completely block the vessels causing a heart attack. This type of disease is the main cause of death worldwide.

Research shows that when the type of plaque causing problems is known, it can help understanding of which narrowing may get worse and cause a heart attack. This information can also help with deciding when and which treatment to provide.

Intravascular imaging is a way to assess the inside of the heart arteries. It involves passing a narrow catheter into the heart vessels. The catheter has a probe on its tip that emits light or an ultrasound signal. The signal is reflected by the vessel wall, back into the probe. A computer program interprets the signals and creates images of the inside of the arteries. There are two types of imaging catheters. One uses sound (Intravascular Ultrasound (IVUS)) and one uses light ((OCT) Optical Coherence Tomography) to produce different types of pictures of the vessels and plaques. The images produced by each type do not provide a full picture of the plaques on their own.

A new hybrid imaging catheter has been developed which has two probes at the tip, an IVUS probe and an OCT probe and can produce both types of images at the same time. It is likely that having both types of images is better for finding high-risk plaques and should lead to better, more specific treatment.

50 heart attack patients who need an angiogram will have images of their vessels taken during their treatment. Once the imaging is complete the patient will continue with their routine planned care.

The information from the images will be used to see how safe and accurate this new hybrid catheter is compared with the separate IVUS and OCT catheters, and also check to see if it is easier to identify plaques that might cause future problems. The study also aims to develop new ways to process and use the images from the hybrid catheter to better treat the plaques that cause the heart attack.

ELIGIBILITY:
Inclusion Criteria:

General Inclusion Criteria

1. Age ≥ 18 to ≤80 years
2. Patient has capacity and willing to consent
3. Must be able to understand English language adequately
4. Patient admitted with an NSTEMI listed for coronary angiography

Angiographic Inclusion Criteria 1) Culprit lesion amenable to PCI

Exclusion Criteria:

General exclusion criteria:

1. eGFR <45ml/min/1.73m²,
2. No known conditions with anticipated life expectancy <1 year,
3. History of heart transplantation,
4. History of Coronary Artery Bypass Grafts (CABG )
5. Intravenous contrast allergy or inability to receive treatment with aspirin, heparin, or thienopyridines,
6. Pregnant or lactating women
7. Decompensated heart failure, or known left ventricular ejection fraction ≤30%

Angiographic exclusion criteria:

1. TIMI 0 flow distally to the culprit lesion,
2. The culprit lesion is located in the left main stem or the ostium of the right coronary artery,
3. Patient that requires surgical revascularization,
4. Unfavourable anatomy for intravascular imaging (i.e., the culprit lesion is a chronic total occlusion or is located in a tortuous vessel where intravascular imaging is not feasible)

Intraprocedural exclusion criteria:

1) If the patient demonstrates evidence of active ischemia or hemodynamic compromise of concern to the operator prior to first insertion of the imaging device (e.g., such as a complication caused by wiring the lesion or after pre-dilating prior to advancing the imaging device for the first time) the study procedure should not commence.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-09-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
To assess the superiority of IVUS-OCT over standalone IVUS in guiding PCI | Measured at procedure
  The number of post PCI findings associated with worse outcomes (i.e., stent un-der expansion, major malappositions, major dissections, large thrombus burden and residual plaque at the edges of the stent) detected by the Conavi Medical Hybrid Imaging System and stand alone IVUS

SECONDARY OUTCOMES:
To examine the safety of the IVUS- OCT catheter in patients undergoing angiography and IVUS-OCT assessment | Measured at procedure, at 1 week post procedure, at 1 month post procedure and 12 months post procedure
  The number of device related complications (vessel perforation, dissection and acute vessel closure during or following IVUS-OCT imaging).
To examine the safety of the IVUS- OCT imaging procedure | Measured at procedure, at 1 week post procedure, at 1 month post procedure and 12 months post procedure
  The number of procedural complications defined as: vessel perforation, angiographic dissection, stent thrombosis, thrombus embolization and acute vessel closure.
To examine the safety of the IVUS- OCT catheter in patients undergoing angiography and intravascular imaging | Measured at procedure, at 1 week post procedure, at 1 month post procedure and 12 months post procedure
  The number of participant deaths or myocardial infarctions

CONTACTS AND LOCATIONS:
Overall Officials: Christos Bourantas, Principal Investigator — Barts & The London NHS Trust
Locations (1):
- St Bartholomew's Hospital, London, England, United Kingdom

IPD SHARING:
Plan to Share IPD: No